CLINICAL TRIAL: NCT03866577
Title: A 4-part Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of M254 in Healthy Volunteers and in Patients With Immune Thrombocytopenic Purpura
Brief Title: Safety and Tolerability of M254 in Healthy Volunteers and Immune Thrombocytopenic Purpura (ITP) Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated based on Sponsor decision.
Sponsor: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108979; 2018-003534-32 (EudraCT Number); MOM-M254-001 (Other: Momenta Pharmaceuticals, Inc.)
Record Dates: First submitted 2019-02-12; First posted 2019-03-07 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Immune Thrombocytopenic Purpura (ITP)
Keywords: Immune thrombocytopenic purpura; Healthy subjects; M254; Intravenous immunoglobulin (IVIg)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Masking Description: Part A: Double (Subject, Investigator);
  Part B, C, and D: Open Label Investigations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A (Experimental): Healthy volunteers will receive a single ascending dose of M254 or placebo
  Interventions: Biological: Biological: M254; Drug: Placebo
- Part B (Experimental): Immune thrombocytopenic purpura (ITP) patients will receive a single ascending dose of M254 followed by IVIg
  Interventions: Biological: Biological: M254; Biological: Intravenous immunoglobulin (IVIg)
- Part C (Experimental): ITP patients will receive a single dose of M254 or IVIg, followed by a single dose of the other drug approximately 28 days later
  Interventions: Biological: Biological: M254; Biological: Intravenous immunoglobulin (IVIg)
- Part D (Experimental): ITP patients will receive repeated doses of M254
  Interventions: Biological: Biological: M254

INTERVENTIONS:
Biological: Biological: M254 — M254 administered as intravenous infusion
Drug: Placebo — Placebo administered as intravenous infusion
  Arms: Part A
Biological: Intravenous immunoglobulin (IVIg) — IVIg administered as intravenous infusion
  Arms: Part B; Part C

SUMMARY:
The purpose of this study is to assess safety, tolerability, pharmacokinetics, and pharmacodynamics of M254 after administration of a single ascending dose and repeat doses in healthy volunteers and immune thrombocytopenic purpura (ITP) patients. The pharmacodynamics of the drug will be measured as platelet response in patients with ITP.

DETAILED DESCRIPTION:
The Part A of the study is currently not accepting healthy volunteers as the recruitment for the part A has completed.

ELIGIBILITY:
Key Criteria for Healthy Volunteers: Subject must be between the ages of 18 and 55 years; healthy as indicated by medical history, physical examination, vital signs, clinical laboratory tests, and 12-lead electrocardiogram, and all abnormal findings are assessed as not clinically significant by the Investigator; not pregnant or breastfeeding; and no other clinically relevant abnormalities currently or in their history that the Investigator would deem them ineligible to participate.

Key Criteria for Immune Thrombocytopenic Purpura (ITP) Patients: Patient must be aged ≥18 years and diagnosed with ITP at least 3 months prior to screening, stable maintenance therapy for at least 4 weeks prior to the first study visit, not pregnant or breastfeeding, and no other clinically relevant abnormalities currently or in their history that the Investigator would deem them ineligible to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Momenta General Queries, Study Director — Momenta Pharmaceuticals, Inc.
Locations (28):
- United States (6):
  - University of Southern California, Los Angeles, California
  - Oncology Institute of Hope and Innovation, Whittier, California
  - Lakes Research, Miami Lakes, Florida
  - University of South Florida, St. Petersburg, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Taussig Cancer Insititute Cleveland Clinic, Cleveland, Ohio
- Ucl de Mont-Godinne, Yvoir, Belgium
- Hungary (3):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Pecsi Tudomanyegyetem, Pécs
- Italy (5):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Azienda Unita Sanitaria Locale di Ravenna, Ravenna
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - Policlinico Universitario Agostino Gemelli, Roma
  - Ospedale 'Casa Sollievo della Sofferenza' - U.O. Ematologia-, San Giovanni Rotondo
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - PRA Health Sciences, Groningen
- Poland (5):
  - Silesian Healthy Blood Clinic, Chorzów
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Szpital Wojewodzki w Opolu, Opole
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej MSW w Poznaniu im prof Ludwika Bierkowskiego, Poznan
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Spain (6):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Burgos, Burgos
  - Hosp. Regional. Carlos Haya, Málaga
  - Hosp. Gral. Univ. J.M. Morales Meseguer, Murcia
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Dr. Peset, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part C Group 2 and Part D of the study was not conducted as planned due to early study termination.
Groups:
- Part A: Pooled Placebo: All healthy participants of Part A received a single intravenous (IV) infusion of matching placebo on Day 1.
- Part A: M254 3 Milligrams/Kilogram (mg/kg): Healthy participants received a single IV infusion of M254 3 mg/kg on Day 1.
- Part A: M254 10 mg/kg: Healthy participants received a single IV infusion of M254 10 mg/kg on Day 1.
- Part A: M254 30 mg/kg: Healthy participants received a single IV infusion of M254 30 mg/kg on Day 1.
- Part A: M254 60 mg/kg: Healthy participants received a single IV infusion of M254 60 mg/kg on Day 1.
- Part A: M254 120 mg/kg: Healthy participants received a single IV infusion of M254 120 mg/kg on Day 1.
- Part A: M254 250 mg/kg: Healthy participants received a single IV infusion of M254 250 mg/kg on Day 1.
- Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg: Participants with immune thrombocytopenia purpura (ITP) received a single IV infusion of M254 20 mg/kg on Day 1 followed by a single IV infusion of IVIg 1000 mg/kg on Day 29.
- Part B: M254 60 mg/kg and IVIg 1000 mg/kg: Participants with ITP received a single IV infusion of M254 60 mg/kg on Day 1 followed by a single IV infusion of IVIg 1000 mg/kg on Day 29.
- Part B: M254 120 mg/kg and IVIg 1000 mg/kg; Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg: Participants with ITP received a single IV infusion of M254 120 mg/kg on Day 1 followed by a single IV infusion of IVIg 1000 mg/kg on Day 29.
- Part B: M254 250 mg/kg and IVIg 1000 mg/kg: Participants with ITP received a single IV infusion of M254 250 mg/kg on Day 1 followed by a single IV infusion of IVIg 1000 mg/kg on Day 29.
- Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg: Participants with ITP received a single IV infusion of IVIg 1000 mg/kg on Day 1 followed by a single IV infusion of M254 120 mg/kg on Day 29.
Period: Overall Study
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg
Started | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 2 | 6 | 5
Completed | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 3 | 2 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Not qualified for IVIg infusion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg | Total
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 2 | 6 | 5 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (10.9) | 31.3 (7.64) | 32 (13.75) | 27 (1) | 29 (7.81) | 32.7 (15.53) | 24.3 (4.51) | 44 (4.24) | 51.8 (11.45) | 44 (12.94) | 54.5 (13.44) | 58 (14.48) | 60 (12.63) | 41.7 (15.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 2 | 0 | 2 | 2 | 1 | 3 | 4 | 1 | 2 | 2 | 26
  Male | 3 | 2 | 1 | 1 | 3 | 1 | 1 | 1 | 2 | 1 | 1 | 4 | 3 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 6 | 1 | 3 | 1 | 3 | 3 | 3 | 2 | 5 | 5 | 2 | 6 | 5 | 45
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Hungary | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 4
  Italy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Netherlands | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 27
  Poland | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 1 | 4 | 2 | 15
  Spain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Parts A, B, and C: Number of Participants With Treatment-emergent Adverse Events (TEAEs) by Severity
Description: An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. A TEAE was defined as any event not present prior to administration of the study drug or any event already present that worsened in either severity or frequency following exposure to the study drug. Severity was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event. Data was planned to be collected and analyzed on pooled population of participants who received placebo in Part A. For Parts B and C, treatment period wise AE data were presented.
Time Frame: From Day 1 up to Day 29
Population: Safety analysis set included all participants who received at least 1 dose of M254 or IVIg or placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: M254 20 mg/kg - M254 Period: Participants with immune thrombocytopenia purpura (ITP) received a single intravenous (IV) infusion of M254 20 mg/kg on Day 1.
- Part B: M254 20 mg/kg - IVIg Period: Participants with ITP received a single IV infusion of IV immunoglobulin (IVIg) 1000 mg/kg on Day 29.
- Part B: M254 60 mg/kg - M254 Period: Participants with ITP received a single IV infusion of M254 60 mg/kg on Day 1.
- Part B: M254 60 mg/kg - IVIg Period; Part B: M254 120 mg/kg - IVIg Period; Part B: M254 250 mg/kg - IVIg Period; Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg - IVIg Period: Participants with ITP received a single IV infusion of IVIg 1000 mg/kg on Day 29.
- Part B: M254 120 mg/kg - M254 Period; Part C (Group 1) : M254 120 mg/kg and IVIg 1000 mg/kg - M254 Period: Participants with ITP received a single IV infusion of M254 120 mg/kg on Day 1.
- Part B: M254 250 mg/kg - M254 Period: Participants with ITP received a single IV infusion of M254 250 mg/kg on Day 1.
- Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg - IVIg Period: Participants with ITP received a single IV infusion of IVIg 1000 mg/kg on Day 1.
- Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg - M254 Period: Participants with ITP received a single IV infusion of M254 120 mg/kg on Day 29.
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg - M254 Period | Part B: M254 20 mg/kg - IVIg Period | Part B: M254 60 mg/kg - M254 Period | Part B: M254 60 mg/kg - IVIg Period | Part B: M254 120 mg/kg - M254 Period | Part B: M254 120 mg/kg - IVIg Period | Part B: M254 250 mg/kg - M254 Period | Part B: M254 250 mg/kg - IVIg Period | Part C (Group 1) : M254 120 mg/kg and IVIg 1000 mg/kg - M254 Period | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg - IVIg Period | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg - IVIg Period | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg - M254 Period
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 5 | 4 | 5 | 3 | 2 | 2 | 6 | 5 | 5 | 5
Participants | 6 | 3 | 3 | 3 | 0 | 3 | 3 | 1 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 2

2. Primary Outcome: Parts A, B, and C: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Values
Description: Number of participants with clinically significant laboratory abnormalities (chemistry, hematology, urinalysis and coagulation) were reported. Data was planned to be collected and analyzed on pooled population of participants who received placebo in Part A.
Time Frame: From Day 1 up to Day 29
Population: Safety analysis set included all participants who received at least 1 dose of M254 or IVIg or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 2 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Parts A, B, and C: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Number of participants with clinically significant abnormalities in vital signs (blood pressure [systolic blood pressure {SBP} and diastolic blood pressure {DBP}], pulse rate, respiratory rate, and body temperature) were reported. Data was planned to be collected and analyzed on pooled population of participants who received placebo in Part A.
Time Frame: From Day 1 up to Day 29
Population: Safety analysis set included all participants who received at least 1 dose of M254 or IVIg or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 2 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Parts A, B, and C: Number of Participants With Clinically Significant Abnormalities in Electrocardiograms (ECGs)
Description: Number of participants with clinically significant abnormalities in ECGs were reported. Data was planned to be collected and analyzed on pooled population of participants who received placebo in Part A.
Time Frame: From Day 1 up to Day 29
Population: Safety analysis set included all participants who received at least 1 dose of M254 or IVIg or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 2 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part C: Maximum Observed Response of M254 (Rmax) on Platelet Count
Description: Rmax is defined as the maximum observed response of M254 on platelet count. Baseline was the pre-dose sample. Data was planned to be collected and analyzed Part C only. For Part C, data were collected and analyzed on the pooled population per the study drug (M254 120 mg/kg and IVIg 1000 mg/kg) which the participants received.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: The full analysis set consisted of all participants who received at least 1 dose of M254 or IVIg or placebo and for whom at least 1 post-infusion pharmacodynamics (PD) assessment was completed. Here, 'N' (number of participants analyzed) indicates number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Groups:
- Part C (Group 1): M254 120 mg/kg - M254 Period (Pooled): Participants with ITP received a single IV infusion of M254 120 mg/kg on Days 1 and 29.
- Part C (Group 1): IVIg 1000 mg/kg - IVIg Period (Pooled): Participants with ITP received a single IV infusion of IVIg 1000 mg/kg on Days 1 and 29.
Arm/Group | Part C (Group 1): M254 120 mg/kg - M254 Period (Pooled) | Part C (Group 1): IVIg 1000 mg/kg - IVIg Period (Pooled)
Number analyzed (Participants) | 11 | 10
10^9 cells per liter | 62.4 (20.1) | 136 (70.0)

6. Primary Outcome: Part C: Change From Baseline in Rmax of M254 in Platelet Count
Description: Change from baseline in Rmax of M254 in platelet count was reported. Rmax is defined as the maximum observed response of M254. Baseline was the predose sample. Therapeutic platelet count was defined as >=50*10^9 cells/L. Platelet response of >=20*10^9 cells/L was considered as increase from baseline. Data was planned to be collected and analyzed for Part C only. For Part C, data were collected and analyzed on the pooled population per the study drug (M254 120 mg/kg and IVIg 1000 mg/kg) which the participants received.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: The full analysis set consisted of all participants who received at least 1 dose of M254 or IVIg or placebo and for whom at least 1 post-infusion PD assessment was completed. Here, 'N' (number of participants analyzed) indicates number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part C (Group 1): M254 120 mg/kg - M254 Period (Pooled) | Part C (Group 1): IVIg 1000 mg/kg - IVIg Period (Pooled)
Number analyzed (Participants) | 11 | 10
10^9 cells per liter | 28.8 (22.2) | 10.5 (67.3)

7. Primary Outcome: Part C: Area Under Effect Curve of the Change From Baseline in Platelet Count From Day 0 to Day 14 (AUEC[0-Day 14]) of M254
Description: AUEC(0-Day 14) is defined as the area under effect curve of the change from baseline in platelet count from Day 0 to Day 14 of M254. Baseline was the predose sample. Data was planned to be collected and analyzed for Part C only. For Part C, data were collected and analyzed on the pooled population per the study drug (M254 120 mg/kg and IVIg 1000 mg/kg) which the participants received.
Time Frame: Predose (baseline) up to Day 14 post dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells *hours per liter
Arm/Group | Part C (Group 1): M254 120 mg/kg - M254 Period (Pooled) | Part C (Group 1): IVIg 1000 mg/kg - IVIg Period (Pooled)
Number analyzed (Participants) | 11 | 10
10^9 cells *hours per liter | 3938 (3952) | 21199 (19349)

8. Primary Outcome: Part C: Area Under Effect Curve of the Change From Baseline in Platelet Count From Day 0 to Day 28 (AUEC[0-Day 28]) of M254
Description: AUEC(0-Day 28) is defined as the area under effect curve of the change from baseline in platelet count from Day 0 to Day 28 of M254. Baseline was the predose sample. Data was planned to be collected and analyzed for Part C only. For Part C, data were collected and analyzed on the pooled population per the study drug (M254 120 mg/kg and IVIg 1000 mg/kg) the participants received.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells *hours per liter
Arm/Group | Part C (Group 1): M254 120 mg/kg - M254 Period (Pooled) | Part C (Group 1): IVIg 1000 mg/kg - IVIg Period (Pooled)
Number analyzed (Participants) | 11 | 10
10^9 cells *hours per liter | 5774 (9453) | 29985 (29265)

9. Secondary Outcome: Part C: Number of Participants With Overall Platelet Response After M254 Administration Compared to IVIg
Description: Number of participants with overall platelet response after M254 administration compared to IVIg were reported. Overall platelet response rate is defined as reaching the therapeutic platelet count. A therapeutic platelet count is defined as greater than or equal to (>=) 50*10^9 cells/liter (L) and an increase from baseline of >=20*10^9 cells/L. Data was planned to be collected and analyzed for Part C only. For Part C, data were collected and analyzed on the pooled population per the study drug (M254 120 mg/kg and IVIg 1000 mg/kg) the participants received.
Time Frame: Up to Day 29
Population: The full analysis set consisted of all participants who were included in the safety set for whom at least 1 post-infusion PD assessment was completed. Here, N (number of participants analyzed) indicates number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Part C (Group 1) : M254 120 mg/kg: Participants with ITP received a single IV infusion of M254 120 mg/kg on Days 1 and 29.
- Part C (Group 1): IVIg 1000 mg/kg: Participants with ITP received a single IV infusion of IVIg 1000 mg/kg on Days 1 and 29.
Arm/Group | Part C (Group 1) : M254 120 mg/kg | Part C (Group 1): IVIg 1000 mg/kg
Number analyzed (Participants) | 11 | 10
Participants | 8 | 9

10. Secondary Outcome: Parts A, B, and C: Maximum Observed Plasma Concentration (Cmax) of M254
Description: Cmax is defined as the maximum observed plasma concentration of M254. Baseline was the predose sample. Data was planned to be collected and analyzed on pooled population of participants who received placebo in Part A. In Part C, combined data of both arms of Group 1 is presented as planned.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: Pharmacokinetic (PK) data analysis set included all randomized participants who received at least 1 dose of M254 or IVIg or placebo with at least 4 evaluable data points adequate to create an evaluable plasma concentration profile of M254.
Measure: Median (Full Range); unit: micrograms per milliliter (mcg/mL)
Groups:
- Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg: Participants with ITP received a single IV infusion of M254 120 mg/kg on Days 1 or 29 and single IV infusion of IVIg 1000 mg/kg on Days 1 or 29.
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 2 | 11
micrograms per milliliter (mcg/mL) | 3.20 [0.600 to 6.10] | 53.9 [51.5 to 55.3] | 174 [172 to 242] | 575 [532 to 664] | 1240 [1148 to 1351] | 2684 [2423 to 3099] | 5444 [3910 to 6316] | 431 [383 to 479] | 1338 [728 to 1724] | 2650 [2480 to 3548] | 5624 [4805 to 6444] | 3068 [2341 to 6008]

11. Secondary Outcome: Parts A, B, and C: Time to Reach Maximum Observed Plasma Concentration (Tmax) of M254
Description: Tmax is defined as the time to reach the maximum observed plasma concentration of M254. Baseline was the predose sample. Data was planned to be collected and analyzed on pooled population of participants who received placebo in Part A. In Part C, combined data of both arms of Group 1 is presented as planned.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: PK data analysis set included all randomized participants who received at least 1 dose of M254 or IVIg or placebo with at least 4 evaluable data points adequate to create an evaluable plasma concentration profile of M254.
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 2 | 11
hours | 338.68 [336.98 to 507.73] | 0.60 [0.60 to 1.10] | 0.45 [0.43 to 2.33] | 0.77 [0.77 to 1.03] | 1.23 [1.20 to 3.18] | 1.83 [1.70 to 2.63] | 2.62 [2.40 to 2.67] | 1.02 [0.87 to 1.17] | 1.48 [1.12 to 1.67] | 1.93 [1.67 to 2.07] | 2.74 [2.53 to 2.95] | 1.85 [1.60 to 2.13]

12. Secondary Outcome: Parts A, B, and C: Area Under the Plasma Concentration-time Curve From Time Zero to Infinite Time (AUC[0-Infinity]) of M254
Description: AUC(0-Infinity) is defined as area under the plasma concentration-time curve from time 0 to infinite time of M254. Baseline was the predose sample. Data was planned to be collected and analyzed on pooled population of participants who received placebo in Part A. In Part C, combined data of both arms of Group 1 is presented as planned.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: PK data analysis set included all randomized participants who received at least 1 dose of M254 or IVIg or placebo with at least 4 evaluable data points adequate to create an evaluable plasma concentration profile of M254. Here, 'N' (number of participants analyzed) indicates number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: micrograms*hour milliliter (mcg*h/mL)
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 1 | 10
micrograms*hour milliliter (mcg*h/mL) | NA [NA to NA] — 'NA' signifies that the median and full range (lower and upper limits) data could not be calculated due to insufficient data available for reliable parameter calculation. | 21488 [12867 to 24589] | 72050 [68012 to 87057] | 210916 [201291 to 223299] | 645641 [521893 to 654506] | 1178098 [997104 to 1351535] | 2196380 [1568703 to 2620469] | 132265 [109746 to 154785] | 423957 [281920 to 527941] | 928888 [847526 to 1000004] | 1839253 [1839253 to 1839253] | 1112165 [693431 to 1377293]

13. Secondary Outcome: Parts A, B, and C: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC[0-Last]) of M254
Description: AUC(0-last) is defined as area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration of M254. AUC(0-last) is calculated by linear-linear trapezoidal summation. Baseline was the predose sample. Data was planned to be collected and analyzed on pooled population of participants who received placebo in Part A. In Part C, combined data of both arms of Group 1 is presented as planned.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: as for outcome 11
Measure: Median (Full Range); unit: mcg*h/mL
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 2 | 11
mcg*h/mL | 593 [52.5 to 1441] | 11531 [9770 to 12701] | 39509 [36176 to 47809] | 111564 [105884 to 121740] | 272532 [251122 to 329379] | 652747 [630464 to 704177] | 1294774 [996669 to 1315203] | 96329 [79956 to 112703] | 287567 [159477 to 415464] | 588913 [546849 to 656664] | 1182466 [1136975 to 1227957] | 700805 [700805 to 1041499]

14. Secondary Outcome: Parts A, B, and C: Apparent Terminal Phase Half-life (t1/2) of M254
Description: t1/2 is defined as the time measured for the plasma concentration to decrease by 1 half to its original concentration of M254. Baseline was the predose sample. Data was planned to be collected and analyzed on pooled population of participants who received placebo in Part A. In Part C, combined data of both arms of Group 1 is presented as planned.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 5 | 1 | 10
hours | NA [NA to NA] — 'NA' signifies that the median and full range (lower and upper limits) data could not be calculated due to insufficient data available for reliable parameter calculation. | 466 [239 to 488] | 463 [412 to 520] | 517 [405 to 530] | 609 [565 to 679] | 659 [468 to 660] | 548 [493 to 762] | 387 [383 to 390] | 478 [427 to 525] | 437 [399 to 595] | 467 [467 to 467] | 391 [254 to 696]

15. Secondary Outcome: Parts A, B, and C: Volume of Distribution (Vz) of M254
Description: Vz is defined as volume of distribution of M254 at terminal phase. Baseline was the predose sample. Data for this outcome measure was not planned for pooled placebo arm in Part A and thus no data was presented for placebo arm in Part A. In Part C, combined data of both arms of Group 1 is presented as planned.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: as for outcome 12
Measure: Median (Full Range); unit: milliliter (mL)
Arm/Group | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 5 | 1 | 10
milliliter (mL) | 6481 [6274 to 7719] | 6129 [5944 to 7396] | 5447 [4445 to 8066] | 7105 [6668 to 7151] | 6383 [4960 to 6468] | 6419 [6087 to 9920] | 8679 [7487 to 9871] | 5259 [5197 to 5321] | 7258 [4907 to 7967] | 9623 [9623 to 9623] | 6059 [2485 to 8707]

16. Secondary Outcome: Parts A, B, and C: Clearance (CL) of M254
Description: CL is defined as clearance of M254, calculated as dose/AUC(0-infinity). Baseline was the predose sample. Data for this outcome measure was not planned for pooled placebo arm in Part A and thus no data was presented for placebo arm in Part A. In Part C, combined data of both arms of Group 1 is presented as planned.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: as for outcome 12
Measure: Median (Full Range); unit: milliliters per hour (mL/h)
Arm/Group | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 5 | 1 | 10
milliliters per hour (mL/h) | 9.63 [8.92 to 22.4] | 9.85 [8.89 to 10.3] | 7.62 [7.30 to 10.5] | 7.59 [7.30 to 8.71] | 6.79 [5.22 to 9.46] | 7.69 [5.84 to 14.0] | 15.6 [13.3 to 17.9] | 12.0 [8.64 to 20.2] | 9.69 [7.79 to 11.7] | 14.3 [14.3 to 14.3] | 10.1 [6.77 to 12.5]

17. Secondary Outcome: Parts A, B, and C: Mean Residence Time (MRT) of M254
Description: Mean residence time is the average time that drug dose remained in the body. Baseline was the predose sample. Data for this outcome measure was not planned for pooled placebo arm in Part A and thus no data was presented for placebo arm in Part A. In Part C, combined data of both arms of Group 1 is presented as planned.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 5 | 1 | 10
hours | 570 (190) | 654 (75.9) | 676 (107) | 867 (79.8) | 820 (163) | 818 (189) | 517 (NA) — 'NA' signifies that the standard deviation was not calculated as planned when the total number of participants analyzed for a treatment was lower than 3. | 661 (77.0) | 653 (109) | 610 (NA) — 'NA' signifies that the standard deviation was not calculated as planned when the total number of participants analyzed for a treatment was lower than 3. | 584 (177)

18. Secondary Outcome: Parts A, B, and C: Percentage of the Estimated Part for the Calculation of AUC(0-infinity) (%AUCextra) of M254
Description: Percentage of the estimated part for the calculation of AUC(0-infinity) (%AUCextra) of M254 were reported. Baseline was the predose sample. Data for this outcome measure was not planned for pooled placebo arm in Part A and thus no data was presented for placebo arm in Part A. In Part C, combined data of both arms of Group 1 is presented as planned.
Time Frame: Predose (baseline) up to Day 29 post dose
Population: PK data analysis set included all randomized participants who received at least 1 dose of M254 or IVIg or placebo with at least 4 evaluable data points adequate to create an evaluable plasma concentration profile of M254. Here, N (number of participants analyzed) indicates number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Percentage of AUC(0-infinity)
Arm/Group | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg and IV Immunoglobulin (IVIg) 1000 mg/kg | Part B: M254 60 mg/kg and IVIg 1000 mg/kg | Part B: M254 120 mg/kg and IVIg 1000 mg/kg | Part B: M254 250 mg/kg and IVIg 1000 mg/kg | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 5 | 1 | 10
Percentage of AUC(0-infinity) | 46.3 [24.1 to 48.3] | 45.1 [41.9 to 49.8] | 49.8 [39.5 to 50.0] | 51.9 [49.7 to 57.8] | 46.5 [34.5 to 47.9] | 40.1 [36.5 to 50.6] | 27.2 [27.1 to 27.2] | 37.0 [31.9 to 43.4] | 31.9 [29.9 to 41.1] | 33.2 [33.2 to 33.2] | 27.6 [17.5 to 50.3]

ADVERSE EVENTS:
Time Frame: From Day 1 up to Day 29
Description: The safety analysis set included all participants who received at least 1 dose of M254 or IVIg or placebo. Data was planned to be collected and analyzed on pooled population of participants who received placebo in Part A. For Parts B and C, treatment period wise AE data were presented.
Groups:
- Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg - M254 Period: Participants with ITP received a single IV infusion of M254 120 mg/kg on Day 1.
Arm/Group | Part A: Pooled Placebo | Part A: M254 3 Milligrams/Kilogram (mg/kg) | Part A: M254 10 mg/kg | Part A: M254 30 mg/kg | Part A: M254 60 mg/kg | Part A: M254 120 mg/kg | Part A: M254 250 mg/kg | Part B: M254 20 mg/kg - M254 Period | Part B: M254 20 mg/kg - IVIg Period | Part B: M254 60 mg/kg - M254 Period | Part B: M254 60 mg/kg - IVIg Period | Part B: M254 120 mg/kg - M254 Period | Part B: M254 120 mg/kg - IVIg Period | Part B: M254 250 mg/kg - M254 Period | Part B: M254 250 mg/kg - IVIg Period | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg - M254 Period | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg - IVIg Period | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg - IVIg Period | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg - M254 Period
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/2 | 0/2 | 0/5 | 0/4 | 0/5 | 0/3 | 0/2 | 0/2 | 0/6 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/2 | 0/2 | 0/5 | 0/4 | 0/5 | 0/3 | 0/2 | 0/2 | 0/6 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 6/7 | 3/3 | 3/3 | 3/3 | 0/3 | 3/3 | 3/3 | 1/2 | 0/2 | 2/5 | 2/4 | 1/5 | 1/3 | 0/2 | 0/2 | 1/6 | 0/5 | 2/5 | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Pooled Placebo (N=7) | Part A: M254 3 Milligrams/Kilogram (mg/kg) (N=3) | Part A: M254 10 mg/kg (N=3) | Part A: M254 30 mg/kg (N=3) | Part A: M254 60 mg/kg (N=3) | Part A: M254 120 mg/kg (N=3) | Part A: M254 250 mg/kg (N=3) | Part B: M254 20 mg/kg - M254 Period (N=2) | Part B: M254 20 mg/kg - IVIg Period (N=2) | Part B: M254 60 mg/kg - M254 Period (N=5) | Part B: M254 60 mg/kg - IVIg Period (N=4) | Part B: M254 120 mg/kg - M254 Period (N=5) | Part B: M254 120 mg/kg - IVIg Period (N=3) | Part B: M254 250 mg/kg - M254 Period (N=2) | Part B: M254 250 mg/kg - IVIg Period (N=2) | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg - M254 Period (N=6) | Part C (Group 1): M254 120 mg/kg and IVIg 1000 mg/kg - IVIg Period (N=5) | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg - IVIg Period (N=5) | Part C (Group 1): IVIg 1000 mg/kg and M254 120 mg/kg - M254 Period (N=5)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces Soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter Site Bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter Site Haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter Site Related Reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling Hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical Device Site Irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel Puncture Site Bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel Puncture Site Haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel Puncture Site Reaction (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Part C (Group 2) and Part D were planned but not conducted based on sponsor decision to discontinue the study after completion of Part A, Part B, and Part C (Group 1). No safety concerns were identified and study was terminated for business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. If this is foreseen, the Investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT03866577/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT03866577/SAP_001.pdf